CLINICAL TRIAL: NCT05546099
Title: Pharmacist-guided, Patient-driven Management of High Blood Pressure in CKD: A Novel Approach
Brief Title: Patient-driven Management of BP in CKD
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIR 21-255
Record Dates: First submitted 2022-09-14; First posted 2022-09-19 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Chronic Kidney Disease
Keywords: kidney disease; hypertension; Home blood pressure; self-management
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Diseases; Hypertension

STUDY DESIGN:
Intervention Model Description: Patients will monitor home BP and adjust meds based on a protocol and under the guidance of a clinical pharmacist.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Self-management (Experimental): Patients monitor their home BP and self manage their BP medications based on a predesigned titration protocol and under the guidance of the clinical pharmacist.
  Interventions: Behavioral: Self-management of BP medications
- Self-monitoring (Active Comparator): Patients monitor their home BP and contact their provider if the BP is above the goal.
  Interventions: Behavioral: Self-monitoring of home BP

INTERVENTIONS:
Behavioral: Self-management of BP medications — Patients will be educated on how to manage their home BP based on a pre-determined protocol. They will then monitor home BP and adjust meds accordingly and under the guidance of the clinical pharmacist.
  Arms: Self-management
Behavioral: Self-monitoring of home BP — Patients will be educated on how to monitor home BP and will be educated to contact their primary care provider/CKD provider if the BP is above the goal.
  Arms: Self-monitoring

SUMMARY:
The proposed research will evaluate if patients managing their blood pressure medications under the guidance of a clinical pharmacist works better to lower blood pressure than patients monitoring their blood pressure at home and the standard care. 60 Veterans with chronic kidney disease (CKD) will be included in the study. The study will further evaluate factors that may influence the Veteran to accept the self-management approach and what factors in the VHA healthcare system affect the implementation of the self-management approach.

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) associates with high morbidity and mortality due to CKD progression and cardiovascular disease (CVD). Blood pressure (BP) lowering reduces the risk of CVD and CKD progression. In spite of the large number of BP medications available, a significant proportion of Veterans with CKD have BP above the goal. The current practice involves licensed providers performing medication titrations to achieve BP goals and is associated with limited patient engagement. The investigators preliminary data indicate that the implementation of pharmacist-guided patient-driven titration of BP medications is effective and feasible in CKD. In this model, Veterans self-manage their BP medications under the guidance of the clinical pharmacist based on a pre-determined medication titration plan.

The prevalence of CKD is extremely high among Veterans, with some studies reporting a prevalence of 47% (vs 11% in the general population). Here, the investigators propose a novel interdisciplinary care model that engages the Veterans as an active participant in their care with the goal of improving BP control to improve long term outcomes. The application addresses a key HSR&D priority (management of complex chronic disease).

The proposed care model is one that has not been tested and includes the clinical pharmacist working with the provider and the Veterans so that Veterans with CKD can self-manage their hypertension. While self-management is exercised in CKD once patients are on dialysis (via home dialysis modalities), the self-management approach is not utilized in the earlier stages of CKD. Importantly, in the approach, the investigators will utilize a transdisciplinary approach to evaluate the implementation of pharmacist-guided self-management of BP medications and the investigators will apply constructs of an implementation science framework, Consolidated Framework for Implementation Research (CFIR), to understand Veteran and system factors that may either facilitate or impede the implementation and sustainment of the pharmacist-guided self-management approach.

Specific aim 1 will evaluate if pharmacist-guided self-management of BP medications is more effective than self-monitoring of home BP + the standard care amongst Veterans with CKD. Specific aim 2 will identify and understand Veteran factors that may influence the acceptability of and the adherence to the self-management approach whereas specific aim 3 will focus on understanding system factors that may facilitate or impede the implementation of the self-management approach.

One hundred and sixty Veterans with uncontrolled hypertension and either stage 2 CKD with albuminuria or stage 3 and 4 CKD will be randomized to either pharmacist-guided self-management or to self-monitoring + the standard practice for 12 months. Aim 1 will evaluate change in [standardized] office systolic BP at 12 months as the primary outcome. Aim 2 will utilize a mixed methods approach including semi-structured interviews to evaluate a sample of 20 Veterans in each of the study arms. The investigators will further design data abstraction tools to evaluate the adherence to the intervention. In aim 3, the investigators will utilize CFIR constructs to guide the investigators qualitative semi-structured interviews with key organizational stakeholders including PACT clinical pharmacists, PCPs, and CKD providers (20 key stakeholders).

The PI will implement the pharmacist-guided self-management approach with the Pharmacy and Ambulatory care services as operational partners. The implementation of this approach will improve the patient experience (Survey of Healthcare Experiences of Patients) and the quality of care (Clinical Performance Measurement Program and the Strategic Analytics for Improvement and Learning).

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years,
* CKD stage 3 or 4 (estimated GFR: 15-59 mL/min/1.73m2) or
* Stage 2 CKD (estimated GFR 60-89 mL/min/1.73m2) with urinary albumin/creatinine ratio (ACR 300 mg/g if no DM and 30 mg/g if with DM), and
* Uncontrolled hypertension defined as the avg of 2 readings > 140 systolic.

Exclusion Criteria:

* Severely uncontrolled hypertension defined as systolic BP >180,
* Patients with resistant hypertension and taking 4 BP medications,
* Orthostatic hypotension defined as reduced systolic BP by 20 mmHg or diastolic BP by 10 mmHg after 3 minutes of standing,
* Severe CKD defined as estimated GFR < 20 mL/min/1.73m2,
* Life expectancy <1 year,
* Severe liver disease,
* Severe congestive heart failure,
* Severe cognitive decline due to dementia,
* Pregnant, breastfeeding, or unwilling to use adequate birth control

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-12-15 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-11-20 (Estimated)

PRIMARY OUTCOMES:
Change in standardized office BP | 12 months
  Detailed procedure for standardized office BP measurement: This will be obtained by a trained research coordinator in accordance with the ACC/AHA and KDIGO (Kidney Disease Improving Global Outcomes) guideline.

SECONDARY OUTCOMES:
Change in conventional office BP | 12 months
  BP measured during standard of care clinical visits will be included.
Home BP readings | 12 months
  The average of the last 10 BP readings at home will be utilized a secondary outcome
Change in standardized office diastolic BP | 12 months
  Measured same as the primary outcome

CONTACTS AND LOCATIONS:
Overall Officials: Diana Jalal, MD, Principal Investigator — Iowa City VA Health Care System, Iowa City, IA
Locations (1):
- Iowa City VA Health Care System, Iowa City, IA, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
Only de- identified research data will be shared with the public. This will only be done under a data use agreement with the requesting entity. A Limited Dataset (LDS) will be created and shared pursuant to a Data Use Agreement (DUA) appropriately limiting use of the dataset and prohibiting the recipient from identifying or re-identifying (or taking steps to identify or re-identify) any individual whose data are included in the dataset.
  If a journal requires that we share the data publicly, then and only then, would we share that data via their requested path. However, no identifiable data, will be shared under any circumstance.
Supporting Information: Study Protocol, SAP
Time Frame: This will be available after the study has concluded, anticipated November 2026 sometime.
Access Criteria: Only de-identified data will be shared via a LDS and only upon request and completion of DUA.

REFERENCES:
- [Derived] Good M, Hoskins R, Lund BC, Ten Eyck P, Dixon B, Cohen J, Reisinger Schact H, Kennelty K, Jalal D. A clinical trial evaluating pharmacist-guided self-management of hypertension among veterans with CKD, rationale and study design. Contemp Clin Trials. 2025 Jul;154:107950. doi: 10.1016/j.cct.2025.107950. Epub 2025 May 11. PMID 40360073